CLINICAL TRIAL: NCT01171768
Title: The Expression of Serum Angiogenesis Marker in Patients Presenting With Hemoptysis
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sang-Won Um, Samsung Medical Center
Other Study IDs: 2008-05-043
Record Dates: First submitted 2010-07-16; First posted 2010-07-28 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Inflammatory Lung Diseases; Hemoptysis
Keywords: Vascular endothelial growth factor; angiopoietin-2
MeSH Terms: conditions — Hemoptysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- patients with hemoptysis within 2 weeks
- patients without hemoptysis within 2 years

SUMMARY:
Vascular endothelial growth factor (VEGF) and angiopoietin-2 (Ang-2) are major mediators of angiogenesis and are induced by tissue inflammation and hypoxia. While elevated serum VEGF levels have been reported in inflammatory lung diseases, especially with hemoptysis, there was no study to evaluate the Ang-2 levels in lung inflammatory diseases according to the presence of hemoptysis, inflammatory biomarker and hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* patients visited Samsung Medical Center for the treatment of benign inflammatory disease such as bronchiectasis, aspergilloma, pneumonia and post-tuberculosis destroyed lung

Exclusion Criteria:

* patients with tumorous condition including lung cancer, vasculitis and the lung disease associated with collagen vascular disease on the point of enrollment

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients visited Samsung Medical Center for the treatment of benign inflammatory disease such as bronchiectasis, aspergilloma, peumonia and post-tuberculosis destroyed lung
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2008-06; Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
serum VEGF and Ang-2 level in lung inflammatory disease according to the presence of hemoptysis | up to 7 days after enrollment
  We'll measure the serum VEFG and Ang-2 level of enrolled patients within a week from the moment that patients agree to enroll this study. Therefore, Comparison of the serum VEGF and Ang-2 level (measured within a week from enrollment) according to the presence of hemoptysis will be primary outcome.

SECONDARY OUTCOMES:
to investigate association between angiogenesis factors and other factors such as inflammatory biomarker and hypoxia. | up to 7 days after enrollment
  We'll measure the serum VEFG, Ang-2 level, and other factors such as inflammatory biomarkers and PaO2 of enrolled patients within a week from the moment that patients agree to enroll this study. Therefore, Investigating association between angiogensis factors and other factors such as inflammatory biomarker and hypoxia, which were measured within a week from enrollment, will be secondary outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea